CLINICAL TRIAL: NCT06757504
Title: A Multi-Center, Randomized, Double-Blind, Parallel Group, Placebo-controlled Phase II Trial of TTYP01 Tablets in Adolescents and Children With Autism Spectrum Disorders
Brief Title: Evaluate the Efficacy and Safety of TTYP01 Tablets in Adolescents and Children With ASD
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Auzone Biological Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TTYP01-Ⅱ-ASD
Record Dates: First submitted 2024-12-25; First posted 2025-01-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder (ASD)
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TTYP01 low-dose group (Experimental): TTYP01 Tablets (12mg or 18mg), Twice daily for 12 weeks. Dosage is determined based on body weight and group assignment, with the low-dose group receiving 12mg-30mg BID, the dosing regimen is detailed in the trial protocol.
  Interventions: Drug: TTYP01 Tablets (12mg or 18mg); Drug: Placebo (Simulant TTYP01 Tablets)
- TTYP01 high-dose group (Experimental): TTYP01 Tablets (12mg or 18mg), Twice daily for 12 weeks. Dosage is determined based on body weight and group assignment, with the high-dose group receiving 24mg-60mg BID, the dosing regimen is detailed in the trial protocol.
  Interventions: Drug: TTYP01 Tablets (12mg or 18mg); Drug: Placebo (Simulant TTYP01 Tablets)
- Placebo group (Placebo Comparator): Simulant TTYP01 Tablets, Twice daily for 12 weeks.
  Interventions: Drug: Placebo (Simulant TTYP01 Tablets)

INTERVENTIONS:
Drug: TTYP01 Tablets (12mg or 18mg) — Taken with a moderate amount of warm water or after disperse in a moderate amount of warm water, at least 60 minutes before breakfast and dinner.
  Arms: TTYP01 high-dose group; TTYP01 low-dose group
Drug: Placebo (Simulant TTYP01 Tablets) — Taken with a moderate amount of warm water or after disperse in a moderate amount of warm water, at least 60 minutes before breakfast and dinner.

SUMMARY:
This is a multi-center, randomized, double-blind, multiple dose levels, parallal group, placebo-controlled study, to evaluate the safety, PK profiles and preliminary efficacy of TTYP01 tablets in adolescents and children with ASD.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, multiple dose levels, parallal group, placebo-controlled study, to evaluate the safety, PK profiles and preliminary efficacy of TTYP01 tablets in adolescents and children with ASD.

The trial will be conducted in 3 stages. It plans to firstly enroll 24 adolescent participants (≥12 to < 16 years) with ASD. After all the 24 adolescent participants have completed the 4-week follow-up and observation, the Data and Safety Monitoring Board (DSMB) will review the data obtained from these adolescent participants, and then make a recommendation on whether to enroll pediatric participants (≥6 to < 12 years) with ASD and continue the adolescent participants' enrollment, whether it is necessary to adjust the protocol, or whether to terminate the trial for safety considerations, etc. If pediatric participants can be enrolled, it plans to first enroll 24 pediatric participants, and the DSMB will review all data after all these participants have completed the 4-week follow-up and observation, and then make a recommendation on whether to continue enrollment of adolescent and pediatric participants, whether to adjust the protocol, or whether to terminate the trial for safety considerations, etc. If the enrollment of adolescent and pediatric participants can be continued, the trial will proceed to Stage 3 until 150 adolescent and pediatric participants with ASD are enrolled. In addition, throughout the trial, the DSMB may conduct irregular reviews of safety, tolerability, PK, and efficacy data, and give recommendations based on the results of the review, including but not limited to adjusting the trial protocol and early termination of the trial for safety considerations. A DSMB review is triggered if a neurotoxicity AE occurs. The composition, responsibilities, etc. of the DSMB are described in Section 4.2 of the protocol.

Eligible participants will be randomized in a 1:1:1 ratio to receive TTYP01 low-dose, TTYP01 high-dose and placebo treatment. Randomization is stratified by age group (≥12 vs < 12 years of age). Participants will be given the corresponding dose of the investigational product for 12 weeks based on their weight and groups as listed in the table in the protocol. The dosing regimen can be adjusted based on the safety, tolerability, PK and other data accumulated in the previous period.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for the study only if all of the following inclusion criteria are met:

1. Aged ≥ 6 to <16 years at the time of signing the ICF (age <16 years after 12-week treatment), including adolescents aged ≥ 12 to<16 years at the time of signing the ICF (age <16 years after 12-week treatment), and children aged ≥ 6 to<12 years at the time of signing the ICF;
2. Male or female;
3. Participants diagnosed with ASD according to the ASD diagnostic criteria in Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) and confirmed by the Schedule for Affective Disorders and Schizophrenia for School Aged Children Present and Lifetime version (K-SADS-PL), DSM-5 ASD module;
4. Child Autism Rating Scale 2-ST (CARS 2-ST) raw score ≥36;
5. CGI-S score ≥4;
6. Participants and their legal guardians understand and are willing to participate in this trial, with ICF signed by the legal guardian and participants aged ≥ 8 years; for participants who, at the discretion of the investigator, have cognitive deficits that prevent them from signing the ICF, their legal guardians sign the ICF on behalf of them;
7. Females of childbearing potential (as defined in Appendix 15.1) agree to remain abstinent or use a reliable method of contraception for the duration of the trial and until 3 months after the last dose of the investigational product.

Exclusion Criteria:

Any participant who meets any of the following criteria will be excluded:

1. Weight <20.0 kg or >70.0 kg, or BMI ≥35.0 kg/m^2;
2. Pregnant or lactating women;
3. Presence of a serious mental disorder as assessed by the investigator, e.g., schizophrenia, bipolar disorder, depressive disorder, etc.; the presence of significant anxiety, tension, agitation, fear, depression, or the presence of suicidal risk, significant risk of self-injury, impulsivity, aggression, or behaviors based on the medical history and the routine mental status examination;
4. History of epileptic seizures within 3 months prior to screening, or presence of a history of severe physical or neurological disease, history of severe head trauma;
5. Participants with a history or symptoms of other mental illness that, at the discretion of the investigator, may affect the results of the study;
6. Participants with a history of any unstable physical or neurological condition or currently suffering from a physical or neurological condition that, at the discretion of the investigator, may put them at risk of a significant adverse event or interfere with the assessment of safety and efficacy during the course of the trial;
7. Pre-existing educational training and/or behavioral treatments fail to be stabilized prior to screening and consistent throughout the trial;
8. Participants who are unable to discontinue or may use other treatments during the screening period and throughout the trial due to their condition, including: antipsychotic medications (except those that may be used in combination during the trial as specified in the protocol), medications that may have a therapeutic effect on ASD, nootropic drugs, medications for ADHD, intestinal flora modification, and other intestinal flora modification supplementation alternatives;
9. Participants who have used treatment modalities such as transcranial magnetic stimulation therapy, direct current stimulation therapy, electroencephalographic biofeedback therapy, auditory integration training, executive function training, acupuncture therapy, etc., within 2 months prior to randomization, or may use such treatments during the treatment period;
10. 12-ECG and laboratory results as outlined below: (1)QTc is outside the normal range of the site; (2)Platelets are below the lower limit of normal for the site; (3)Haemoglobin is below the lower limit of normal for the site; (4)Neutrophil count is below the lower limit of normal for the site; (5)ALT or AST ≥ 2 × upper limit of normal, or total bilirubin > upper limit of normal for the site; (6)Urea nitrogen or creatinine is above the upper limit of normal for the site; (7)Any other abnormal laboratory, vital sign, or 12-ECG findings that, at the discretion of the investigator, are abnormal and clinically significant and will affect the safety of the participant or the interpretation of the study results;
11. Participation in any clinical trial of a drug or non-drug intervention within the last 1 month;
12. Concomitant medications/therapies that are prohibited in the protocol may be required during the trial;
13. Participants expected to undergo elective surgery during the trial;
14. Participants whose parents/guardians are unable to understand and/or complete the scale assessments in this trial.
15. Hypersensitivity to edaravone and excipients (Soluplus, sodium bisulphite, microcrystalline cellulose, magnesium stearate, polyvinylpolypyrrolidone) in TTYP01 tablets;
16. Participants who are judged by the investigator to be ineligible for other reasons.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in ABC-SW（Aberrant Behavioral Checklist - Social Withdrawal） scores at Week 12. | At baseline and week 12
  The ABC (Aberrant Behavioral Checklist) scale has 58 items. The scale is broken down into five subscales including ABC-SW（Aberrant Behavioral Checklist - Social Withdrawal）, ABC-I, A, C （Aberrant Behavioral Checklist - Irritability, Agitation, Crying）, ABC-SB （Aberrant Behavioral Checklist - Stereotypic Behavior）, ABC-H, N (Aberrant Behavioral Checklist - Hyperactivity, Noncompliance ), and ABC-IS (Aberrant Behavioral Checklist - Inappropriate Speech ). Scale ratings can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others with knowledge of the person being assessed.
  The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Incidence and severity of treatment-emergent adverse events (TEAEs), adverse events of special interest (AESIs), serious adverse events (SAEs), and TEAEs that lead to treatment discontinuation. | Throughout the trial period
  To evaluate the safety and tolerability of TTYP01 tablets in adolescent and pediatric participants with ASD.
Plasma concentrations and population PK profiles of edaravone and its metabolites in adolescent and pediatric ASD participants. | Visit 2 (Day 1): 30 minutes (±5 minutes) and 3 hours (±10 minutes) after the first dose; Visit 8 (Week 12 ±2 Days)or Early withdrawal: before the first dose (0 hour), and 30 minutes (±5 minutes) after the first dose on the day of the visit.
  Concentrations of edaravone and its metabolites are assayed in the plasma of adolescent and pediatric participants with ASD. They will be analyzed with descriptive statistics according to planned sampling points.

SECONDARY OUTCOMES:
Changes from baseline in ABC-SW scores at Weeks 4 and 8. | At baseline, Weeks 4 and 8
  The ABC (Aberrant Behavioral Checklist) scale has 58 items. The scale is broken down into five subscales including ABC-SW（Aberrant Behavioral Checklist - Social Withdrawal）, ABC-I, A, C （Aberrant Behavioral Checklist - Irritability, Agitation, Crying）, ABC-SB （Aberrant Behavioral Checklist - Stereotypic Behavior）, ABC-H, N (Aberrant Behavioral Checklist - Hyperactivity, Noncompliance ), and ABC-IS (Aberrant Behavioral Checklist - Inappropriate Speech ). Scale ratings can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others with knowledge of the person being assessed.
  The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Changes from baseline in other ABC subscale scores at Weeks 4, 8 and 12. | At baseline, Weeks 4, 8 and 12
  The ABC (Aberrant Behavioral Checklist) scale has 58 items. The scale is broken down into five subscales including ABC-SW（Aberrant Behavioral Checklist - Social Withdrawal）, ABC-I, A, C （Aberrant Behavioral Checklist - Irritability, Agitation, Crying）, ABC-SB （Aberrant Behavioral Checklist - Stereotypic Behavior）, ABC-H, N (Aberrant Behavioral Checklist - Hyperactivity, Noncompliance ), and ABC-IS (Aberrant Behavioral Checklist - Inappropriate Speech ). Scale ratings can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others with knowledge of the person being assessed.
  The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Clinical Global Impressions-Improvement (CGI-I) scores at Weeks 4, 8, and 12. | At Weeks 4, 8, and 12.
  The CGI includes the CGI-S and CGI-I. The CGI rating scale allows for an overall assessment of participant improvement over time. At baseline, the CGI-S assessment is performed and the rating investigator rates the severity of the participant's condition based on a 7-point scale ranging from 1 (no symptoms) to 7 (very severe symptoms). At the follow-up visit, the scoring investigator assessed the degree of improvement in the participant's symptoms relative to baseline based on the CGI-I items on a 7-point scale ranging from 1 (very marked improvement) to 7 (very marked deterioration).
Changes from baseline in Clinical Global Impressions-Severity (CGI-S) scores at Weeks 4, 8, and 12. | At baseline, Weeks 4, 8 and 12
  The CGI includes the CGI-S and CGI-I. The CGI rating scale allows for an overall assessment of participant improvement over time. At baseline, the CGI-S assessment is performed and the rating investigator rates the severity of the participant's condition based on a 7-point scale ranging from 1 (no symptoms) to 7 (very severe symptoms). At the follow-up visit, the scoring investigator assessed the degree of improvement in the participant's symptoms relative to baseline based on the CGI-I items on a 7-point scale ranging from 1 (very marked improvement) to 7 (very marked deterioration).
Changes from baseline in Social Responsiveness Scale 2 (SRS-2) total scores at Weeks 4, 8, and 12. | At baseline, Weeks 4, 8 and 12
  The SRS-2 assesses participants' social communication, social awareness, social motivation, and self-regulation. Scales can be completed by parents and teachers.Both the SRS-2 total score and the five subscale scores can be used to assess the severity of ASD symptoms. The SRS-2-School Age was used in this study.
  The SRS-2 contains 65 items, each of which is rated by the assessor on a scale of 1 (not true), 2 (sometimes true), 3 (often true), and 4 (almost always true) based on the behavioral performance of the person being assessed. Scores range from 65-260, where higher scores indicate more severe social problems.
Changes from baseline in Autism Treatment Evaluation Checklist (ATEC) total scores at Weeks 4, 8, and 12. | At baseline, Weeks 4, 8 and 12
  The ATEC contains four subscales: language/communication, social, sensory/cognitive awareness, and health/physical/behavioral, and scale ratings can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others who know the person being assessed.
  Scores from each subscale are combined to calculate a total score, which ranges from 0 to 179. Higher scores indicate more severe autism symptoms and behavioral problems, and lower scores indicate improvement in symptoms.
Changes from baseline in the total score of the Attention-Deficit Hyperactivity Disorder Rating Scale-IV - Home version (ADHD-RS-IV [Home version]) at Weeks 4, 8, and 12. | At baseline, Weeks 4, 8 and 12
  The ADHD-RS assesses the child's attention deficit and hyperactive/impulsive behaviors over the past six months. Scale ratings can be completed by parents and teachers.
  The ADHD-RS consists of 18 items that cover various aspects of attention and hyperactivity symptoms. Participants assess the extent of each item based on their performance using a four-point scale:0 (Never or Rarely), 1 (Sometimes), 2 (Often), and 3 (Very Often). By combining these items, a composite score can be derived that measures the severity of attention deficit and hyperactivity symptoms. Higher scores indicate more severe symptoms.
Changes from baseline in Behavior Rating Inventory of Executive Function (BRIEF) (Parent Version) scores at Weeks 4, 8, and 12. | At baseline, Weeks 4, 8 and 12
  The Children's BRIEF (Parent Version) assesses executive functioning in children and adolescents, including aspects of working memory, planning/organization, and task monitoring, and the scale can be completed by a parent or guardian. The first version of the Children's BRIEF (Parent Version) was used in this study.
  The parent version of the BRIEF for school-age children assesses the executive functioning of children aged 6 to 18 years old, and contains 86 items divided into 2 latitudes: behavioral regulation index (BRI, including 3 factors of inhibition, switching and emotional control) and metacognition index (MI, including 5 factors of task initiation, working memory, planning, organizing and monitoring). Each item was rated on a scale of 1 to 3 (1=never; 2=sometimes; 3=often), with higher ratings reflecting more severe impairment of executive function.
Proportion of participants with ≥25% reduction in ABC-SW score relative to baseline at Week 12. | At baseline and week 12
  The ABC (Aberrant Behavioral Checklist) scale has 58 items. The scale is broken down into five subscales including ABC-SW（Aberrant Behavioral Checklist - Social Withdrawal）, ABC-I, A, C （Aberrant Behavioral Checklist - Irritability, Agitation, Crying）, ABC-SB （Aberrant Behavioral Checklist - Stereotypic Behavior）, ABC-H, N (Aberrant Behavioral Checklist - Hyperactivity, Noncompliance ), and ABC-IS (Aberrant Behavioral Checklist - Inappropriate Speech ). Scale ratings can be completed by parents, special educators, psychologists, direct caregivers, nurses, and others with knowledge of the person being assessed.
  The rater has to answer each of the 58 questions using a 4-point Likert scale. A score of a "0" means the behavior is not a problem, a score of a "1" means slight problem, a score of a "2" means a serious problem, and a "3" means a severe problem.
Proportion of participants with a CGI-I score ≤ 2 at Week 12. | At Week 12
  The CGI includes the CGI-S and CGI-I. The CGI rating scale allows for an overall assessment of participant improvement over time. At baseline, the CGI-S assessment is performed and the rating investigator rates the severity of the participant's condition based on a 7-point scale ranging from 1 (no symptoms) to 7 (very severe symptoms). At the follow-up visit, the scoring investigator assessed the degree of improvement in the participant's symptoms relative to baseline based on the CGI-I items on a 7-point scale ranging from 1 (very marked improvement) to 7 (very marked deterioration).

OTHER OUTCOMES:
Changes from baseline in the proportion of time spent looking at different facial areas and social situations in eye-tracking tasks by eye-tracking method at Week 12 of administration. | At baseline and week 12
  Exploratory objective metrics that may predict benefit from TTYP01 tablets
Changes from baseline in fNIRS examination at Week 12. | At baseline and week 12
  Exploratory Outcomes, Objectivity indicators that may predict benefit from TTYP01 tablets
Changes from baseline in the level of plasma cytokines (i.e., IL-1β, IL-6, TNF-α, INF-γ, IL-7, IL-12, and IL-17) at Week 12. | At baseline and week 12
  Exploratory Outcomes, Biomarker indicators that may predict benefit from TTYP01 tablets
Changes from baseline in the levels of plasma reduced glutathione (GSH), oxidized glutathione (GSSG), and GSH/GSSG at Week 12. | At baseline and week 12
  Exploratory Outcomes, Biomarker indicators that may predict benefit from TTYP01 tablets
Changes from baseline in Total Antioxidant Capacity (T-AOC) of urine at Week 12. | At baseline and week 12
  Exploratory Outcomes, Biomarker indicators that may predict benefit from TTYP01 tablets

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, Study Chair — Peking University Sixth Hospital
Locations (5):
- China (5):
  - Peking University Sixth Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Nanjing Brain Hospital, The Affiliated Brain Hospital of Nanjing Medical University, Nanjing
  - Tianjin Mental Health Center, Tianjin